CLINICAL TRIAL: NCT06534021
Title: A Phase Ia Study to the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of IASO-782 in Patient With Autoimmune Hematological Diseases (Autoimmune Thrombocytopenia and Warm Antibody Type Autoimmune Hemolytic Anemia)
Brief Title: IASO-782 in Autoimmune Hematological Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai IASO Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IASO-782C005
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Autoimmune Thrombocytopenia; Warm Autoimmune Haemolytic Anaemia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Drug:IASO-782 injection Dosage and Administration: single dose of IASO-782, 6 mg/kg or 10 mg/kg , intravenous injection at day 1
  Interventions: Drug: IASO-782 injection
- Control group (Placebo Comparator): Drug:placebo Dosage and Administration: single dose of placebo, intravenous injection at day 1
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IASO-782 injection — Each subject will be given only one dose of IASO-782. Subjects should avoid strenuous exercise within 48 h before administration and remain seated or semi-recumbent (except for necessary activities) for 4 h after administration. IASO-782 solution for injection or placebo was diluted in 0.9% sodium chloride injection (corresponding to the dose administered according to the body weight at baseline and the dose group) with a total volume of 250 mL, administered as a single intravenous drip at a drip rate recommended by the drug manual on the day of administration, The infusion time is about 90 minutes (± 15 minutes).
  Arms: Experimental group
Drug: placebo — Each subject will be given one dose of placebo. Subjects should avoid strenuous exercise within 48 h before administration and remain seated or semi-recumbent (except for necessary activities) for 4 h after administration. IASO-782 solution for injection or placebo was diluted in 0.9% sodium chloride injection (corresponding to the dose administered according to the body weight at baseline and the dose group) with a total volume of 250 mL, administered as a single intravenous drip at a drip rate recommended by the drug manual on the day of administration, The infusion time is about 90 minutes (± 15 minutes).
  Arms: Control group

SUMMARY:
This study is a randomized, double-blinded, and placebo-controlled phase Ia clinical study in subjects with autoimmune hematological diseases. The study is designed to assess the safety and tolerability of IASO-782 for the treatment of autoimmune haematological diseases (ITP and wAIHA).

DETAILED DESCRIPTION:
This study is a single-dose escalation study in subjects with autoimmune hematological diseases. The study is designed to enroll subjects with autoimmune thrombocytopenia and warm antibody type immune haemolytic anaemia (ITP and wAIHA).

Referred to the clinical pharmacological study and development experience of similar drugs, one or more dose regimens will be determined for the use in Phase 1b clinical trials.

This study will evaluate the safety and preliminary dose range of IASO-782 in subjects with autoimmune hematologic diseases (ITP and wAIHA) at the following dose levels:6mg/kg and 10mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Clinically confirmed diagnosis of autoimmune thrombocytopenia (ITP) or warm autoimmune haemolytic anaemia (wAIHA)
3. Failure or relapse after at least 1 treatment for the study disease
4. Stable dose of immunosuppressants for 4 weeks before screening
5. Organ function or laboratory test is basically normal
6. Subjects of childbearing potential and their partners must use effective contraception for at least 2 weeks before administration of investigational product, throughout the trial period, and for 28 days after the end of the trial (or early termination of the trial)
7. Females of potential childbearing capacity must have a negative pregnancy test at screening
8. Voluntarily participate in this study and sign the informed consent

Exclusion Criteria:

1. History of other primary malignant neoplasm within 5 years of screening
2. Secondary to other disease-induced hematopoietic destruction
3. Cardiac disorder within the last 3 months
4. Patients with high blood pressure that cannot be controlled by drug
5. Subjects with a history of allergy to any component of the investigational drug
6. Active infection requiring intravenous treatment within 30 days prior to the enrollment
7. Pregnant or breastfeeding women
8. Participation was being given other investigational drug within 30 days or 5 half-lives (whichever is longer) prior to administration of the investigational drug
9. Previous treatment drugs have not been adequately washed out
10. ITP patients have had any previous arterial or venous thrombosis
11. Patients with ITP had previous biopsy bone marrow results indicating bone marrow fibrosis (Myelofibrosis MF) ≥ 2
12. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C (HCV) infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection, as described in the protocol
13. Subjects with a history of drug abuse or mental disorder
14. Other medical history or conditions that would make the subject unsuitable for the study by investigators' judge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0 | up to 12 weeks
  The safety and tolerability of IASO-782 will be assessed primarily by summarizing treatment-emergent AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No